CLINICAL TRIAL: NCT04669548
Title: Physiologic Signals and Signatures With the Accuryn Monitoring System - A Retrospective and Prospective Analysis (The Accuryn Registry)
Brief Title: Physiologic Signals and Signatures With the Accuryn Monitoring System - The Accuryn Registry
Status: Recruiting | Type: Observational
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-06-101904
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Intraabdominal Hypertension; Abdominal Compartment Syndrome; Acute Kidney Injury; Cardiovascular Surgery
Keywords: Acute Kidney Injury (AKI); CABG; Cardiovascular Surgery; Intraabdominal Pressure (IAP); Urine Output (UO); Accuryn
MeSH Terms: conditions — Intra-Abdominal Hypertension; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Accuryn Monitoring System: Observational only (no intervention). Patients undergoing cardiovascular surgical intervention(s) monitored with the Accuryn Monitoring System (per standard of care) during their hospital stay
  Interventions: Device: Accuryn Monitoring System

INTERVENTIONS:
Device: Accuryn Monitoring System — The Accuryn Monitoring System is a novel Foley catheter and monitoring device capable of detecting physiologic changes in vital signs via sensors within the catheter system. These data are captured non-invasively, continuously, and at a high frequency.

SUMMARY:
The Accuryn Registry Study is an open-ended, global, multi-center, retrospective and prospective, single-arm data collection study with an FDA cleared device. The target population are cardiovascular surgery patients. Physiologic data measurements will be collected from enrolled subjects using electronic medical records and data streams via the Accuryn Monitoring System.

DETAILED DESCRIPTION:
The primary objective of the Accuryn Registry Study is to is to track and analyze changes in physiologic data streams using the Accuryn Monitoring System and correlate these changes to the occurrence of acute kidney injury (AKI) following cardiac surgical intervention(s).

The secondary objective is to determine the incidence of intraoperative and postoperative intra-abdominal hypertension in the cardiovascular surgery population, analyze what factors may contribute to the development of intra-abdominal hypertension (IAH) in this patient population, and analyze associations of IAH with organ dysfunctions such as acute kidney injury and other clinical outcomes (e.g. ICU length of stay, required hemodialysis, readmission).

ELIGIBILITY:
Inclusion Criteria:

1. Signed or Verbal Informed Consent as required by IRB (if applicable).
2. Adult (age ≥ 18).
3. Monitored on the Accuryn® Monitoring System during their procedure and ICU stay (for retrospective enrollment).
4. Patient is undergoing cardiac surgical intervention(s).

Exclusion Criteria:

1. Known history of advanced chronic kidney disease defined by an estimated glomerular filtration rate (eGFR) <20 mL/min/1.73m2 within 30 days prior to procedure.
2. The patient is unsuitable for the study, in the opinion of the investigator. This may include vulnerable patient populations such as pregnant women, prisoners ,or those detained in a penal institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiovascular surgical intervention(s) who meet eligibility criteria and are monitored with the Accuryn Monitoring System throughout their procedure and intensive care unit (ICU) stay.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Urine Output (UO) | 30 days
  High accuracy Urine Output (mL/hour) while on a urinary catheter, and estimated UO while not on a urinary catheter
Intra-Abdominal Pressure (IAP) | 30 days
  Intra-Abdominal Pressure (mmHg) trending while on a urinary catheter, as well as active measurements taken by clinician clinician
Temperature (T) | 30 days
  Temperature (degrees Celsius) trending during hospital stay
Intraabdominal Hypertension (IAH) | 30 days
  Intra-abdominal pressure (IAP) above 12 mm Hg (timepoint and duration)
Abdominal Compartment Syndrome (ACS) | 30 days
  Intra-abdominal pressure (IAP) above 20 mm Hg with new organ dysfunction or failure (timepoint and duration)
Acute Kidney Injury (AKI) | 30 days
  % of patients diagnosed with AKI, and hospitalization day of diagnosis. AKI diagnosed per KDIGO criteria (Stage 1 to 3)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Moll, MD, PhD, Study Director — Potrero Medical
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - San Francisco VA Medical Center, San Francisco, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Jewish Hospital / University of Louisville, Louisville, Kentucky
  - Mission Health Hospital, Asheville, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khanna AK, Minear S, Kurz A, Moll V, Stanton K, Essakalli L, Prabhakar A; Predict AKI Group. Intra-abdominal hypertension in cardiac surgery patients: a multicenter observational sub-study of the Accuryn registry. J Clin Monit Comput. 2023 Feb;37(1):189-199. doi: 10.1007/s10877-022-00878-2. Epub 2022 Jun 13. PMID 35695943